CLINICAL TRIAL: NCT03000816
Title: A Phase 2 Study of Stereotactic Body Radiotherapy (SBRT) for the Treatment of OligoMetastatic Esophageal Squamous Cell Carcinoma
Brief Title: A Study of SBRT for OligoMetastatic ESCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESO-Shanghai10
Record Dates: First submitted 2016-12-18; First posted 2016-12-22 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Esophageal Squamous Cell Carcinoma Metastatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental Arm (Experimental): Patients in this arm will receive a treatment of SBRT for their oligometastatic lesions.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Patients with 1-4 metastases located in less than 2 organs/ lymphatic drainage regions that are 5 cm or less from each other and simultaneously treated with SBRT.

SUMMARY:
The aim of this phase II trial is to assess progress-free survival, local control, overall survival, safety and tolerability of SBRT to treat patients with oligometastases in esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with metastatic esophageal squamous cell carcinoma who have received initial treatment for the primary site including surgery or chemoradiotherapy. Primary tumor site without progression at registration. The sites of allowed metastases are: peripheral lung, central lung, medistinal/cervical lymph node, liver, spinal/paraspinal, osseous, and abdominal-pelvic lymph node. All metastases not resected must be amenable to SBRT.
2. 1-4 radiographically distinct metastases of any distribution in 2 or less allowed anatomical sites. The diameters of lesions should be less than or equal to 5cm.
3. Initial treatment should be completed at least 3 months prior to study registration.
4. All the metastases treated with SBRT should not be treated with surgery, radiation, radio frequency ablation or other regional therapeutic modalities prior to study registration. The other (s) lesions should have been surgically removed.
5. Age ≥ 18. PS ECOG 0-2，wight loss<30% during the latest 6 months.
6. Evaluation by a radiation oncologist that the patient could tolerate the treatment of SBRT.
7. Patient must provide study specific informed consent prior to study entry.
8. For females of child-bearing potential, negative serum/urine pregnancy test within 14 days prior to study registration.

Exclusion Criteria:

1. Progression of primary tumor site at time of registration.
2. Metastases with indistinct borders making targeting not feasible.
3. Known brain metastases.
4. Prior palliative radiotherapy to metastases.
5. Metastases located within 3 cm of the previously irradiated structures:

   a).Spinal cord previously irradiated >80Gy(Biological equivalent dose with α/β=2), b).Brachial plexus previously irradiated to > 100Gy(Biological equivalent dose with α/β=2), c).Small intestine, large intestine, or stomach previously irradiated to > 90Gy (Biological equivalent dose with α/β=2), d).Whole lung previously irradiated with prior V20Gy > 30% (delivered in ≤ 3 Gy/fraction), e)Metastasis irradiated with SBRT.
6. Pregnant or breast-feeding women or people during the birth-period who refused to take contraceptives.
7. Drug addiction,Alcoholism or AIDS.
8. Patients with severe organ dysfunction or Acute bacterial or fungal infection who are considered not suitable to enroll the study at the time of registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | The survival time from the date each patient enrolled to the date of progression or date of death from any cause, whichever came first, assessed up to 5 years
  progression-free survival will be measured as time to either progression or death

SECONDARY OUTCOMES:
Local control | the time from the date each patient enrolled to the date of local failure or the last follow-up, assessed up to 5 years.
  Local control will be measured as time to local recurrence
overall survival | The survival time from the date each patient enrolled to the date of death or the last follow-up, assessed up to 5 years.
  Overall survival will be measured as time until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Kuaile Zhao, MD., Study Chair — Fudan Universtiy Shanghai Cancer Center
Locations (1):
- Fudan Universtiy Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Q, Zhu Z, Chen Y, Deng J, Ai D, Liu Q, Wang S, Wu S, Chen J, Zhao K. Phase 2 Study of Stereotactic Body Radiation Therapy for Patients with Oligometastatic Esophageal Squamous Cell Carcinoma. Int J Radiat Oncol Biol Phys. 2020 Nov 1;108(3):707-715. doi: 10.1016/j.ijrobp.2020.05.003. Epub 2020 May 14. PMID 32417405